CLINICAL TRIAL: NCT05490420
Title: Effects of Upper Extremity Manual Lymphatic Drainage on Symptom Severity, Hand Functions, Electrophysiological and Ultrasonographic Measurements in Carpal Tunnel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Emel Mete, research assistant, Istanbul Medeniyet University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/0344
Record Dates: First submitted 2022-08-04; First posted 2022-08-05 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2022-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; manual lymphatic drainage; surface electromyography
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Manual Lymphatic Drainage

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: participant will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): 17 participants who meet the inclusion criteria will be applied conventional exercise which includes nerve gliding and tendon gliding exercises. And also sham (placebo) upper extremity manual lymphatic drainage will be applied. Sham (placebo) manual lymphatic drainage will include only classical massage not manual lymphatic drainage techniques. Participants will be treated for a total of 6 weeks, 2 days a week. Each session will last approximately 20-30 minutes, and the exercises will be performed in 3 sets with 10 repetitions.
  Interventions: Other: manual lymphatic drainage (MLD)
- experimental (Experimental): 17 participants who meet the inclusion criteria will be applied both conventional exercise and upper manual lymphatic drainage (MLD). MLD is a manual technique that is applied to the lymphatic system with a pressure of approximately 40-50mmHg and increases the working speed of lymphatic nodules/collectors. Its main purpose is to support microcirculation by accelerating lymphatic flow and to prevent/remove interstitial fluid accumulation that may cause fascial adhesions. Within the scope of this research, an application will be made to cover the entire upper extremity lymphatic system. MLD will last approximately 20-30 minutes. Conventional exercise, which includes nerve gliding and tendon gliding exercises, will be performed in 3 sets with 10 repetitions. Participants will be treated for a total of 6 weeks, 2 days a week.
  Interventions: Other: manual lymphatic drainage (MLD)

INTERVENTIONS:
Other: manual lymphatic drainage (MLD) — MLD is a manual technique that is applied to the lymphatic system with a pressure of approximately 40-50mmHg and increases the working speed of lymphatic nodules/collectors. Its main purpose is to support microcirculation by accelerating lymphatic flow and to prevent/remove interstitial fluid accumulation that may cause fascial adhesions.

SUMMARY:
This study is aimed to investigate the effects of upper extremity manual lymphatic drainage, which is applied to remove edema from the carpal tunnel region in addition to conventional exercise therapy in Carpal tunnel syndrome patients on findings of clinical, ultrasonographic, and electrophysiological.

DETAILED DESCRIPTION:
Thirtyfour volunteer participants between aged 40 and 60 years, who met the inclusion criteria, will be included in the study. Participants will be randomly divided into two groups experimental and control groups. While the control group will receive only conventional exercises, the experimental group will receive both conventional exercises and upper extremity manual lymphatic drainage. A total of 3 measurements will be made before the treatment, after the treatment and 1 month after the end of the treatment. Symptom severity will be evaluated via Boston carpal tunnel syndrome questionnaire, grip strength via hand dynamometer, pressure pain threshold via digital algometer device, cross-sectional area of the median nerve via ultrasound, and median nerve conduction velocity via superficial EMG device.

ELIGIBILITY:
Inclusion Criteria:

* People aged between 40-60 years
* Having been diagnosed with carpal tunnel syndrome (CTS) at least 6 months ago or having symptoms related to carpal tunnel syndrome for at least 6 months
* Having mild (median nerve sensory conduction velocity below 40 m/sec) and moderate (median nerve sensory conduction velocity below 40 m/sec and median motor distal latency 4 ms and above) CTS according to electrophysiological findings
* Not having received medical treatment and/or physiotherapy for CTS in the last 6 months

Exclusion Criteria:

* Having cervical radiculopathy
* Having thoracic outlet syndrome
* Presence of systemic disease that may lead to CTS, such as diabetes or thyroid disease
* Pregnancy
* Presence of anemia
* Having a history of CTS surgery
* Presence of radial or ulnar nerve sensory-motor lesions accompanying the present condition
* Presence of lymphedema
* Having severe (Sensory nerve action potential cannot be obtained) and severe (Sensory nerve action potential cannot be obtained, but combined muscle action potential is not present) CTS according to electrophysiological findings

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2022-09-05 (Actual); Primary Completion 2023-06-03 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Symptom severity | Change from baseline symptom severity at week 6 and 10.
  1- Symptom severity will be evaulated with Boston carpal tunnel questionnaire (BCTQ). BCTQ comprises 11 items of Symptom Severity Scale (SSS) measuring pain, paresthesia, numbness, nocturnal symptoms and feeling of weakness plus another 8 items of Functional Status Scale (FSS) measuring difficulties in performing daily activities. Scales ranged from 1-5 representing normal to worst symptoms or disabilities. Higher scores indicate greater symptom severity and disability.
Grip strength | Change from baseline grip strength at week 6 and 10.
  2- Grip strength will be assessed with a digital hand dynamometer. The subject will seat with feet positioned on the floor, shoulder adducted, and the elbow bent at a 90-degree angle with the forearm parallel to the floor. Maximal isometric grip strength will be measured in kilograms. It is a reliable method for measuring grip strength.
Pressure pain threshold (PPT) | Change from baseline pressure pain threshold at week 6 and 10.
  PPT, the minimal amount of pressure where a sense of pressure changes to pain, will be measured with an electronic algometer over the median nerve in the wrist area. The pressure will be applied approximately at a rate of 30 kPa/sec for 30 seconds. Participants will be instructed to press the switch when the sensation changed from pressure to pain.
Cross-sectional area of the median nerve | Change from baseline cross-sectional area of the median nerve at week 6 and 10.
  US images will be obtained by a neurologist trained in peripheral nerve US. The nerve will be imaged using a Biosound Esaote MyLab 70 equipped with an 18-MHZ linear-array transducer. The median nerve will be imaged in cross-section at the distal wrist crease (carpal tunnel inlet) and 12 cm proximal to this point in the forearm.
Sensory Velocity of median nerve | Change from baseline Sensory Velocity of median nerve at week 6 and 10.
  Sensory Velocity of median nerve will be recorded with surface EMG using surface electrodes from the abductor pollicis brevis (APB) muscle by a neurologist using standard techniques.
Motor velocity of median nerve | Change from baseline motor velocity of median nerve at week 6 and 10.
  Motor Velocity of median nerve will be recorded with surface EMG using surface electrodes from the abductor pollicis brevis (APB) muscle by a neurologist using standard techniques

CONTACTS AND LOCATIONS:
Locations (1):
- Emel Mete, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided